CLINICAL TRIAL: NCT04019041
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Bermekimab in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of Bermekimab in Patients With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108834; 77474462HDS2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa; Suppurative Hidradenitis
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — bermekimab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to every week bermekimab injections, every other week bermekimab injections, or every week placebo injections.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- bermekimab ew (Experimental): 2 800 mg bermekimab loading dose subcutaneous injections, followed by weekly 400 mg bermekimab injections
  Interventions: Drug: bermekimab
- bermekimab eow (Experimental): 2 800 mg loading dose subcutaneous injections, followed by alternating weekly 400 mg bermekimab injections with matching placebo injections
  Interventions: Drug: bermekimab; Drug: placebo
- placebo ew (Placebo Comparator): 2 800 mg placebo loading dose subcutaneous injections, followed by weekly placebo subcutaneous injections
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bermekimab — bermekimab 2 mL (200 mg/mL) pre-filled syringe
  Arms: bermekimab eow; bermekimab ew
Drug: placebo — placebo 2 mL pre-filled syringe
  Arms: bermekimab eow; placebo ew

SUMMARY:
This study further evaluates the efficacy of bermekimab in treating moderate to severe hidradenitis suppurativa in adults. 1/3 of patients will receive weekly injections of bermekimab, 1/3 will receive alternating every other week injections of bermekimab or placebo, and 1/3 will receive weekly injections of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the participant
* Male or female, age greater than or equal to (>=) 18 years
* Naïve to OR failure of prior targeted biologic therapy for Hidradenitis Suppurativa (HS) (including anti-TNF, anti-IL-17, or JAK inhibitor therapy)
* Diagnosis of HS for at least 1 year prior to screening.
* HS affecting at least two distinct anatomic areas, one of which is Hurley II or III stage.
* A total body count of abscesses and inflammatory nodules (AN) of at least 3.
* Full understanding of the procedures of the study protocol and willingness to comply with them.
* In case of female participants of childbearing potential, willingness to use one method of contraception of high efficacy during the entire study period. This method can be hormonal contraceptives or one of the following: condoms, diaphragm, or an intrauterine device. Women of non-childbearing potential include those considered to have a medical history that indicates that pregnancy is not a reasonable risk, including post-menopausal women and those with a history of hysterectomy or surgically sterilized.

Exclusion Criteria:

* Age below 18 years.
* History of treatment with bermekimab for any reason.
* Receipt of oral antibiotic treatment for HS within 28 days prior to baseline.
* Receipt of prescription topical therapies for the treatment of HS within 14 days prior to baseline, and/or systemic non-biologic therapies for HS (immunosuppressants, corticosteroids, retinoids, or hormonal therapies) within 28 days prior to screening.
* Participant has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to baseline.
* History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies.
* Has received a live (attenuated) vaccine over the 28 days prior to screening.
* Participant received oral concomitant analgesics (including opioids) for HS-related pain within 14 days prior to baseline.
* If entering the study on concomitant oral analgesics (including opioids) for non-HS-related pain: (a) Participant on opioid analgesics within 14 days prior to baseline visit; (b) Participant not on a stable dose of non-opioid oral analgesics for at least 14 days prior to baseline visit (PRN is not considered a stable dose).
* Participant requires or is expected to require opioid analgesics for any reason (excluding tramadol).
* Participant has a draining fistula count of greater than 20 at baseline.
* Major surgery (requiring general anesthesia or respiratory assistance) within 28 days prior to Day 0 of start of study drug.
* Hepatic dysfunction defined as any value of transaminases, of γ-glutamyl transpeptidase (γGT) or of total bilirubin > 3x upper normal limit.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution.
* Stage C Child-Pugh liver cirrhosis.
* History of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Neutropenia defined as <1,000 neutrophils/mm3.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (33):
- United States (33):
  - Desert Sky, Gilbert, Arizona
  - Marvel Clinical Research, Huntington Beach, California
  - University of Southern California, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Syrentis Clinical Research, Santa Ana, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Visionary Investigators Network, Aventura, Florida
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Doral Medical Research, Doral, Florida
  - Floridian Research Institute, Miami, Florida
  - Florida International Medical Research, Miami, Florida
  - P&S Research, LLC, Miami, Florida
  - Accel Clinical Research, Orlando, Florida
  - Physica Clinical Research, Sebastian, Florida
  - Avita Clinical Research, Tampa, Florida
  - Forcare Clinical Research, Inc., Tampa, Florida
  - Integrated Clincal Research LLC, West Palm Beach, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Randall Dermatology & Cosmetic Surgery, West Lafayette, Indiana
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Clinical Trials of SWLA, Lake Charles, Louisiana
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - ClinOhio Research Services, Columbus, Ohio
  - Clinical Research Solutions, LLC, Milan, Tennessee
  - Progressive Clinical Research, San Antonio, Texas
  - Dominion Medical Associates, Inc., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Week 0-16): Participants received placebo as subcutaneous (SC) injection at Weeks 0 and 1, and once every week (qw) from Week 2 through Week 16.
- Bermekimab 400 mg q2w (Week 0-16): Participants received loading dose of bermekimab 800 milligrams (mg) (2*400 mg) as SC injection at Weeks 0 and 1, followed by bermekimab 400 mg once every 2 weeks (q2w) alternating with matching placebo q2w through Week 16.
- Bermekimab 400 mg qw (Week 0-16): Participants received loading dose of bermekimab 800 mg (2*400 mg) as SC injection at Weeks 0 and 1, followed by bermekimab 400 mg qw through Week 16.
- Placebo to Bermekimab 400 mg qw (Week 17-36): At Week 16, participants who received placebo during placebo-controlled period entered into active treatment period and received bermekimab 400 mg as SC injection qw through Week 31. All participants entered safety follow-up (F-u) at Week 32 through Week 36.
- Bermekimab 400 mg q2w (Week 17-36): At Week 16, participants who received bermekimab 400 mg q2w during placebo-controlled period entered into active treatment period and received bermekimab 400 mg as SC injection q2w with matching placebo through Week 31. All participants entered safety follow-up at Week 32 through Week 36.
- Bermekimab 400 mg qw (Week 17-36): At Week 16, participants who received bermekimab 400 mg qw during placebo-controlled period entered into active treatment period and continued to receive bermekimab 400 mg as SC injection qw through Week 31. All participants entered safety follow-up at Week 32 through Week 36.
Period: Placebo Controlled Period (Weeks 0-16)
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16) | Placebo to Bermekimab 400 mg qw (Week 17-36) | Bermekimab 400 mg q2w (Week 17-36) | Bermekimab 400 mg qw (Week 17-36)
Started | 52 | 50 | 51 | 0 | 0 | 0
Completed | 48 | 43 | 43 | 0 | 0 | 0
Not Completed | 4 | 7 | 8 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Imprisonment/compulsory detention | 0 | 0 | 1 | 0 | 0 | 0
Period: Active Treatment+Safety F-U (Week 17-36)
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16) | Placebo to Bermekimab 400 mg qw (Week 17-36) | Bermekimab 400 mg q2w (Week 17-36) | Bermekimab 400 mg qw (Week 17-36)
Started | 0 | 0 | 0 | 48 | 43 | 43
Completed | 0 | 0 | 0 | 42 | 35 | 38
Not Completed | 0 | 0 | 0 | 6 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16) | Total
Number analyzed (Participants) | 52 | 50 | 51 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 45 | 48 | 143
  >=65 years | 2 | 5 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13.65) | 37.2 (13.85) | 40.4 (14.02) | 38.9 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 41 | 37 | 113
  Male | 17 | 9 | 14 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 1 | 0 | 0 | 1
  Black or African American | 14 | 16 | 13 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 33 | 33 | 33 | 99
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
  Other | 3 | 1 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 52 | 50 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR was defined as at least 50 percent (%) reduction in total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 12
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
Percentage of participants | 46.2 | 44.0 | 54.9

2. Secondary Outcome: Change From Baseline in Numeric Rating Scale (NRS) for Pain & Itch at Weeks 12 and 16
Description: Change from baseline in NRS for pain and itch at Weeks 12 and 16 was reported. Participants were given a take-home diary to complete each night before bed. Participants were asked to report "average pain", and "worst moment pain" as well as "average itch" and "worst moment itch" on a 0 to 10 NRS, where 0=no itch or no pain and 10=worst itch or worst pain. Higher score indicated more severity.
Time Frame: Baseline, Week 12, Week 16
Population: The FAS included all randomized participants who received at least 1 dose of study agent. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 41 | 44 | 41
scores on a scale
  Pain: Week 12: number analyzed (Participants) | 40 | 44 | 41
  Pain: Week 12 | -1.47 (1.987) | -1.92 (2.528) | -1.67 (2.472)
  Pain: Week 16 | -1.52 (2.086) | -1.80 (2.537) | -1.63 (2.307)
  Itch: Week 12: number analyzed (Participants) | 40 | 44 | 41
  Itch: Week 12 | -1.79 (2.356) | -1.82 (2.767) | -1.62 (2.764)
  Itch: Week 16 | -1.66 (3.081) | -1.29 (2.940) | -1.45 (2.660)

3. Secondary Outcome: Change Form Baseline in Total Abscess and Inflammatory Nodule (AN) Count at Weeks 12 and 16
Description: Change form baseline in total AN count at Weeks 12 and 16 was reported. Abscess and inflammatory nodule were counted for the hidradenitis suppurativa (HS) affected anatomical regions. The AN count is the sum of number of abscess and inflammatory nodules across anatomical regions.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Abscess and inflammatory nodule
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 49 | 46 | 47
Abscess and inflammatory nodule
  Week 12 | -3.7 (7.95) | -4.0 (6.97) | -5.2 (6.18)
  Week 16: number analyzed (Participants) | 48 | 46 | 47
  Week 16 | -5.1 (8.11) | -4.8 (8.31) | -5.1 (6.54)

4. Secondary Outcome: Change From Baseline in Number of Draining Fistulas at Weeks 12 and 16
Description: Change form baseline in number of draining fistulas at Weeks 12 and 16 was reported. Draining fistula were defined as fistulas that drain serious or purulent fluid, either spontaneously or by gentle palpation.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: fistulas
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 49 | 46 | 47
fistulas
  Week 12 | -0.6 (1.90) | 0.1 (4.54) | -0.3 (0.82)
  Week 16: number analyzed (Participants) | 48 | 46 | 47
  Week 16 | -0.6 (2.56) | -0.5 (1.17) | -0.3 (1.76)

5. Secondary Outcome: Percentage of Participants Who Achieved Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: HiSCR was defined as at least 50% reduction in AN count with no increase in abscess count and no increase in draining fistula count relative to baseline.
Time Frame: Week 16
Population: The FAS included all randomized participants who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
percentage of participants | 44.2 | 52.0 | 56.9

6. Secondary Outcome: Change From Baseline in Modified Hidradenitis Suppurativa Score (mHSS) at Weeks 12 and 16
Description: Change from baseline in mHSS at Weeks 12 and 16 was reported. The sartorius scale was used to quantify the severity of HS. Points were awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other): points were awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); other findings (1 point); and longest distance between 2 lesions (2-6 points, 0 if no lesions); and if lesions were separated by normal skin (yes: 0 points; no: 6 points). The total sartorius score was the sum of the 12 regional scores. Scale scores range from 0 to infinite, with larger scores representing higher severity of HS.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 49 | 46 | 47
scores on a scale
  Week 12 | -24.0 (35.36) | -13.2 (42.54) | -26.1 (20.94)
  Week 16: number analyzed (Participants) | 48 | 46 | 47
  Week 16 | -26.8 (43.19) | -22.4 (44.53) | -24.1 (30.47)

7. Secondary Outcome: Percentage of Participants Who Achieved HS-PGA of Clear (0) or Minimal (1) or HS-PGA Score of Mild or Better (<=2) With at Least a 2-grade Improvement Relative to Baseline at Weeks 12 and 16
Description: HS-PGA was physician assessment of severity of disease based on 6-point scale:Clear (0)=total number of abscesses, inflammatory nodule, non-inflammatory nodule and draining fistulas was 0;Minimal (1)=total number of abscesses,draining fistulas, inflammatory nodule was 0, presence of non-inflammatory nodule;Mild (2)=total number of abscesses, draining fistulas was 0, total number of inflammatory nodule was 1-4, or presence of 1 abscess or draining fistula and absence of any inflammatory nodules;Moderate (3)=total number of abscesses and draining fistulas was 0, total number of inflammatory nodule was at least 5; or presence of 1 abscess or draining fistula and at least 1 inflammatory nodule; or 2-5 abscesses or draining fistulas, fewer than 10 inflammatory nodule;Severe (4)=total number of abscesses or draining fistulas was 2-5, total number of inflammatory nodule was at least 10;Very severe (5)=more than 5 abscesses or draining fistulas.Higher score indicated more severity of disease.
Time Frame: Weeks 12 and 16
Population: The FAS included all randomized participants who received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
percentage of participants
  Week 12 | 11.5 | 2.0 | 17.6
  Week 16 | 11.5 | 2.0 | 19.6

8. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score at Weeks 12 and 16
Description: The HADS was an instrument for screening anxiety and depression in non-psychiatric populations; repeated administration also provides information about changes in a participant's emotional state. It comprises 14 items, seven to assess anxiety (HADS-A), namely items 1, 3, 5, 7, 9, 11, and 13; and seven to assess depression (HADS-D), namely items 2, 4, 6, 8, 10, 12, and 14. Each item receives a score from 0 to 3 on a Likert Scale. The total score for each HADS-A and HADS-D scale was obtained by adding the individual scores for each item, with the maximum score 21. The presence or absence of depression and anxiety was defined, for each respective scale, based on the following cutoff values: HADS (anxiety): 0-8 equal to (=) no anxiety; greater than (>) 9 = anxiety; HADS (depression): 0-8 = no depression; >9 = depression.
Time Frame: Baseline, Week 12, Week 16
Population: The FAS included all randomized participants who received at least 1 dose of study agent. Here, 'n' (number analyzed) signifies participants who were evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
scores on a scale
  HADS anxiety: Week 12: number analyzed (Participants) | 51 | 49 | 49
  HADS anxiety: Week 12 | -1.7 (2.70) | -1.4 (3.54) | -1.5 (3.65)
  HADS anxiety: Week 16 | -1.6 (3.19) | -1.8 (3.17) | -1.8 (3.13)
  HADS depression: Week 12: number analyzed (Participants) | 51 | 49 | 49
  HADS depression: Week 12 | -0.6 (2.58) | -0.8 (2.41) | -1.5 (3.48)
  HADS depression: Week 16 | -0.5 (2.43) | -0.9 (2.53) | -1.3 (3.15)

9. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Weeks 12 and 16
Description: DLQI was a simple, compact, and practical questionnaire to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. The DLQI domains include symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The participant respond on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best. A lower score (that is, negative change score) indicated improvement in the Quality of Life.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 50
scores on a scale
  Week 12: number analyzed (Participants) | 50 | 49 | 49
  Week 12 | -3.8 (4.91) | -4.5 (7.09) | -4.6 (5.07)
  Week 16 | -4.2 (5.92) | -5.1 (7.09) | -4.7 (5.27)

10. Secondary Outcome: Change From Baseline in Health Status as Assessed by EuroQol-5 Dimension Instrument-3 Levels (EQ-5D-3L) Visual Analogue Scale (VAS) Scores at Weeks 12 and 16
Description: The EQ-5D-3L was a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It consists of EQ-5D descriptive system and EQ visual analogue scale (VAS). EQ-5D-3L-VAS records the participant's self-rated health on a vertical VAS that allows the participants to indicate their health state that can range from 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicated improvement.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
scores on a scale
  Week 12: number analyzed (Participants) | 51 | 49 | 50
  Week 12 | 7.2 (14.30) | 6.9 (14.69) | 3.7 (19.20)
  Week 16 | 9.3 (14.23) | 7.7 (14.60) | 6.1 (17.47)

11. Secondary Outcome: Number of Participants With Patient Global Impression of Change (PGI-c) at Week 12 and 16
Description: The PGI-c was a single-item patient reported outcome (PRO) that assessed change in severity of skin pain due to HS. Participants rated how his/her HS had changed since the beginning of the study using a 7-point scale ranging from 1 to 7 where 1 indicates "very much better", 2 indicates "Much better', 3 indicates "A little better", 4 indicates "No change", 5 indicates "A little worse", 6 indicates "Much worse" and 7 indicates "Very much worse".
Time Frame: Week 12, Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 48 | 42 | 44
Participants
  Very much better: Week 12: number analyzed (Participants) | 47 | 41 | 44
  Very much better: Week 12 | 3 | 1 | 7
  Much better: Week 12: number analyzed (Participants) | 47 | 41 | 44
  Much better: Week 12 | 6 | 3 | 5
  A little better: Week 12: number analyzed (Participants) | 47 | 41 | 44
  A little better: Week 12 | 5 | 14 | 6
  No change: Week 12: number analyzed (Participants) | 47 | 41 | 44
  No change: Week 12 | 14 | 14 | 15
  A little worse: Week 12: number analyzed (Participants) | 47 | 41 | 44
  A little worse: Week 12 | 13 | 6 | 8
  Much worse: Week 12: number analyzed (Participants) | 47 | 41 | 44
  Much worse: Week 12 | 5 | 3 | 2
  Very much worse: Week 12: number analyzed (Participants) | 47 | 41 | 44
  Very much worse: Week 12 | 1 | 0 | 1
  Very much better: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Very much better: Week 16 | 4 | 1 | 6
  Much better: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Much better: Week 16 | 9 | 6 | 3
  A little better: Week 16: number analyzed (Participants) | 48 | 42 | 43
  A little better: Week 16 | 7 | 8 | 12
  No change: Week 16: number analyzed (Participants) | 48 | 42 | 43
  No change: Week 16 | 13 | 17 | 12
  A little worse: Week 16: number analyzed (Participants) | 48 | 42 | 43
  A little worse: Week 16 | 12 | 6 | 7
  Much worse: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Much worse: Week 16 | 2 | 4 | 2
  Very much worse: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Very much worse: Week 16 | 1 | 0 | 1

12. Secondary Outcome: Number of Participants With Patient Global Impression of Severity (PGI-s) at Weeks 12 and 16
Description: The PGI-s was a single-item PRO that assessed change in a participant's impression of their disease severity. The PGI-s item asks the respondent to best describe how his/her HS symptoms are now (that is, "check the one number that best describes how your HS symptoms are now") on a 4-point scale scored as: "normal" (1), "mild" (2), "moderate" (3), or "severe" (4)".
Time Frame: Week 12, Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 48 | 42 | 44
Participants
  Normal: Week 12: number analyzed (Participants) | 46 | 41 | 44
  Normal: Week 12 | 7 | 3 | 7
  Mild: Week 12: number analyzed (Participants) | 46 | 41 | 44
  Mild: Week 12 | 12 | 19 | 19
  Moderate: Week 12: number analyzed (Participants) | 46 | 41 | 44
  Moderate: Week 12 | 15 | 19 | 14
  Severe: Week 12: number analyzed (Participants) | 46 | 41 | 44
  Severe: Week 12 | 12 | 0 | 4
  Normal: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Normal: Week 16 | 7 | 3 | 8
  Mild: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Mild: Week 16 | 18 | 22 | 16
  Moderate: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Moderate: Week 16 | 13 | 15 | 11
  Severe: Week 16: number analyzed (Participants) | 48 | 42 | 43
  Severe: Week 16 | 10 | 2 | 8

13. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa (HS)-Related Pain Symptom Score in the Past 24 Hours Based on Hidradenitis Suppurativa Symptom Diary (HSSD) Questionnaire at Weeks 12 and 16
Description: HSSD is a 7-item patient self-reported questionnaire that assesses 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms have a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours with a score range from 0 (no symptom experience) to 10 (worst possible symptom experience). A total symptom score also ranged from 0 (no symptom) to 10 (worst possible symptom), was derived by averaging the 5 individual scale scores that utilize the past 7-day recall period. Change from baseline in HS-related pain symptom score in the past 24 hours based on HSSD was reported.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 51 | 50 | 50
scores on a scale
  Week 12: number analyzed (Participants) | 51 | 49 | 50
  Week 12 | -1.7 (2.81) | -1.8 (3.05) | -1.9 (2.81)
  Week 16 | -1.9 (2.83) | -1.9 (2.97) | -1.9 (2.85)

14. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa Symptom Diary (HSSD) Total Symptom Score at Weeks 12 and 16
Description: The HSSD was a 7-item patient self-reported questionnaire that assessed 5 HS-related symptoms including pain, tenderness, hot skin feeling, odor, and itchiness. The participants were asked to rate the severity of each symptom on a 0 to 10 numerical rating scale, with 0 indicating no symptom experience and 10 indicating the worst possible symptom experience. All 5 symptoms had a recall period of the past 7 days, except for 2 additional questions on pain which evaluate current pain and pain in the past 24 hours. Each individual symptom scale score, ranging from 0-10, was summarized. A total symptom score, which also ranged from 0-10, was derived by averaging the 5 individual scale scores that utilize the past 7-day recall period.
Time Frame: Baseline, Week 12, Week 16
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 52 | 50 | 51
scores on a scale
  Week 12: number analyzed (Participants) | 51 | 49 | 50
  Week 12 | -1.9 (2.16) | -2.1 (2.38) | -2.1 (2.19)
  Week 16 | -1.8 (2.01) | -2.0 (2.33) | -1.9 (2.29)

15. Secondary Outcome: Serum Concentration of Bermekimab
Description: Serum concentration of bermekimab was reported. This outcome measure was planned to be analyzed for specified arms only.
Time Frame: Baseline (Week 0), Weeks 1, 2, 3, 4, 5, 8, 12, and 16
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 complete dose of bermekimab and had at least 1 valid blood sample drawn for PK analysis after their first dose of bermekimab. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies participants who were evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 50 | 50
micrograms per milliliter (mcg/mL)
  Week 0 | 0.00 (0.000) | 0.00 (0.000)
  Week 1: number analyzed (Participants) | 47 | 47
  Week 1 | 31.60 (18.697) | 35.76 (19.153)
  Week 2: number analyzed (Participants) | 43 | 46
  Week 2 | 37.75 (20.620) | 48.81 (25.938)
  Week 3: number analyzed (Participants) | 42 | 47
  Week 3 | 16.44 (12.725) | 38.09 (25.627)
  Week 4: number analyzed (Participants) | 42 | 44
  Week 4 | 20.22 (14.118) | 34.71 (21.042)
  Week 5: number analyzed (Participants) | 38 | 43
  Week 5 | 9.94 (9.794) | 30.95 (20.248)
  Week 8: number analyzed (Participants) | 34 | 38
  Week 8 | 21.43 (15.529) | 28.34 (17.659)
  Week 12: number analyzed (Participants) | 26 | 31
  Week 12 | 20.87 (13.407) | 29.36 (16.891)
  Week 16: number analyzed (Participants) | 28 | 32
  Week 16 | 21.35 (17.958) | 31.03 (18.503)

16. Secondary Outcome: Reduction From Baseline in Serum Interleukin-6 (IL-6)
Description: Reduction from baseline in serum IL-6 was reported.
Time Frame: Baseline, Weeks 8, 12 and 16
Population: Due to change in planned analysis, data was not collected for this outcome measure hence analysis was not performed.
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Placebo Controlled Period: Weeks 0 to 16; Active Treatment + Safety Follow-up Period: Weeks 17 to 36
Description: The safety analysis set included all randomized participants who received at least 1 dose of study agent, that is, the treated population.
Arm/Group | Placebo (Week 0-16) | Bermekimab 400 mg q2w (Week 0-16) | Bermekimab 400 mg qw (Week 0-16) | Placebo to Bermekimab 400 mg qw (Week 17-36) | Bermekimab 400 mg q2w (Week 17-36) | Bermekimab 400 mg qw (Week 17-36)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/51 | 0/48 | 1/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/52 | 0/50 | 1/51 | 0/48 | 3/43 | 2/43
Other Adverse Events (participants affected / at risk) | 16/52 | 14/50 | 13/51 | 10/48 | 4/43 | 6/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=52) | Bermekimab 400 mg q2w (Week 0-16) (N=50) | Bermekimab 400 mg qw (Week 0-16) (N=51) | Placebo to Bermekimab 400 mg qw (Week 17-36) (N=48) | Bermekimab 400 mg q2w (Week 17-36) (N=43) | Bermekimab 400 mg qw (Week 17-36) (N=43)
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 0-16) (N=52) | Bermekimab 400 mg q2w (Week 0-16) (N=50) | Bermekimab 400 mg qw (Week 0-16) (N=51) | Placebo to Bermekimab 400 mg qw (Week 17-36) (N=48) | Bermekimab 400 mg q2w (Week 17-36) (N=43) | Bermekimab 400 mg qw (Week 17-36) (N=43)
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 2 | 4 | 3 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 2 | 1 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 1 | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 2 | 2 | 1 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 4 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04019041/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04019041/SAP_001.pdf